CLINICAL TRIAL: NCT02371837
Title: Effects of 6 Week of Pilates in Fall Prevention
Brief Title: Effects of Pilates in Risk Fall in Older Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Professor., University of Jaén
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UJA2015
Record Dates: First submitted 2015-02-09; First posted 2015-02-26 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Falling Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pilates group (Experimental): Pilates based protocol for 6 weeks
  Interventions: Other: Pilates and fall prevention
- control group (No Intervention): No treatment group

INTERVENTIONS:
Other: Pilates and fall prevention — A 2 days per week during 6 week Pilates practice will be performed in experimental group in order to check the effectiveness in fall prevention
  Arms: pilates group

SUMMARY:
The intervention will consist in a 6 week of pilates practice in older population to check the prevention of fall effectiveness.

DETAILED DESCRIPTION:
A study population of elder people will be randomly allocated to intervention or control group, consisted in Pilates and a booklet of balance tips respectively.

The protocol will be performed for 6 weeks.

ELIGIBILITY:
Inclusion Criteria: - Elder population. Not to be a pilates practitioner previous to study enrollment. Exclusion Criteria: - Cognitive issues that dont allow to practice pilates method.

Sensorial alteration or any disease that could altered balance. Any drug or medication that modify balance.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Falls Efficacy Scale International test (FES I) | pre intervention and post 6 weeks of intervention
  FES as measure of fear of falling or patients confident of falling

SECONDARY OUTCOMES:
Change in Star Excursion Balance Test (SEBT) | pre intervention and post 6 weeks of intervention
  SEBT as measure of dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Martinez, PhD, Principal Investigator — IBIMER University of Granada
Locations (1):
- University of Jaén, Jaén, Andalusia, Spain